CLINICAL TRIAL: NCT02121340
Title: Collaborative Care for Depression and Diabetic Retinopathy in African Americans
Acronym: CC-DDR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Wills Eye (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34EY024299 (NIH)
Record Dates: First submitted 2014-04-21; First posted 2014-04-23 (Estimated); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Diabetic Retinopathy
Keywords: Depression; Health disparities; African American; Geriatric
MeSH Terms: conditions — Diabetic Retinopathy; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavioral Activation (Experimental): CC-DDR is a novel mental health/ophthalmologic intervention that we are designing to treat depression and lower HbA1C levels in older AAs with mild-to-moderate DR and comorbid depression. Community Health Workers, who match participants in race and cultural background, will work with ophthalmologists in the retina clinic to educate participants on the links between depression, HbA1C, and DR, and will extend care into the home where they will use Behavioral Activation to treat depression and improve diabetes self-management skills.
  Interventions: Behavioral: Behavioral Activation
- Usual Care (No Intervention): Usual Care

INTERVENTIONS:
Behavioral: Behavioral Activation
  Arms: Behavioral Activation

SUMMARY:
In this feasibility/pilot study, we will develop, refine, and evaluate the feasibility of a novel mental health/ophthalmologic intervention called, "Collaborative Care for Depression and Diabetic Retinopathy" (CC-DDR), which aims to treat depression and lower HbA1C in older African Americans with mild-to-moderate diabetic retinopathy (DR) and comorbid depression.

DETAILED DESCRIPTION:
The Specific Aims are:

1. To develop the CC-DDR treatment protocol. This will involve:

   1. Creating an initial version of the CC-DDR treatment protocol.
   2. Refining the protocol based on input from an expert panel with expertise in DR, depression, and culturally relevant interventions for diabetes in older African Americans.
   3. Developing a tool to assess interventionist treatment adherence and competence.
2. To conduct an open trial of CC-DDR with 40 participants who have poorly controlled diabetes, depression, and mild or moderate DR. During this open trial we will:

   1. Evaluate the feasibility of CC-DDR.
   2. Refine the CC-DDR treatment protocol by incorporating feedback from participants, community health care workers (CHWs), ophthalmologists, and the expert panel.
   3. Refine procedures for recruitment and retention, outcome assessment, monitoring treatment fidelity, CHW training and supervision, quality assurance, and study administration, based on input from investigators, CHWs, participants, and the expert panel.
   4. Examine CC-DDR's impact on depression severity; diabetes self-management practices; HbA1C level; blood pressure; adherence to the ophthalmologist treatment plan; vision function; quality of life; and satisfaction with CC-DDR.
3. To complete a Manual of Procedures that characterizes all aspects of the planned efficacy trial of CC-DDR.

ELIGIBILITY:
Inclusion Criteria:

1. African-American race
2. age ≥ 65 years
3. type 2 diabetes
4. mild or moderate nonproliferative DR with or without macular edema
5. depressive symptoms (i.e., Patient Health Questionnaire-9 score ≥5)
6. HbA1C ≥ 7.0%

Exclusion Criteria:

1. treated proliferative DR
2. global cognitive impairment (i.e., Mini Mental Status score ≤ 20)
3. psychiatric diagnosis other than depression
4. treatment for depression started in the previous 3 months
5. life expectancy under 2 years

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-05 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | 12 months
  Change in hemoglobin A1c from baseline to 12 months

OTHER OUTCOMES:
Depression | 12 months
  Improvement in depressive symptoms from baseline to 12 months
Progression of diabetic retinopathy | Baseline to 12 months
Diabetes self management | 12 months
  Improvement from baseline to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Barry Rovner, MD, Principal Investigator — Thomas Jefferson University; Robin Casten, PhD, Study Director — Thomas Jefferson University
Locations (2):
- United States (2):
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Wills Eye Hospital, Philadelphia, Pennsylvania